CLINICAL TRIAL: NCT00072930
Title: Phase II, Randomized, Open-Label, Two-Arm, Multicenter Study of MEDI-522, a HuMA Directed Against the Human Alpha V Beta 3 Integrin, in Combination With Docetaxel, Prednisone, and Zoledronic Acid in the Treatment of Patients With Metastatic Androgen-Independent Prostate Cancer
Brief Title: MEDI-522 in the Treatment of Patients With Metastatic Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Luz Hammershaimb, M.D., V.P., Clinical Dev., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP098
Record Dates: First submitted 2003-11-12; First posted 2003-11-17 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — etaracizumab; Docetaxel; Prednisone; Zoledronic Acid

ARMS (2):
- 1 (Active Comparator): MEDI-522 + Docetaxel + Prednisone + Zoledronic Acid (N=55)
  Interventions: Biological: MEDI-522
- 2 (Other): Docetaxel + Prednisone + Zoledronic Acid (N=55)
  Interventions: Biological: Docetaxel + Prednisone* + Zoledronic Acid

INTERVENTIONS:
Biological: MEDI-522 — IV at a concentration of 50 mg/mL and 10mL vials
  Arms: 1
Biological: Docetaxel + Prednisone* + Zoledronic Acid — IV 75 mg/m2 IV 3-4 mg 5 mg
  Arms: 2

SUMMARY:
The primary objectives of this study are:

1. To explore the antitumor activity of MEDI-522 in combination with docetaxel, prednisone, and zoledronic acid in patients with metastatic Androgen-Independent Prostate Cancer (AIPC); and
2. To summarize the safety of MEDI-522 in combination with docetaxel, prednisone, and zoledronic acid in this patient population.

DETAILED DESCRIPTION:
This is a Phase II, randomized, open-label, two-arm, multicenter study of MEDI-522 in combination with docetaxel, prednisone, and zoledronic acid in patients with metastatic AIPC.

ELIGIBILITY:
Inclusion Criteria:

* Adult men at least 18 years of age at the time of randomization.
* Metastatic, histologically or cytologically confirmed adenocarcinoma of the prostate that has progressed after start of androgen deprivation therapy, which includes prior orchiectomy or medical castration using leuteinizing hormone-releasing hormone (LHRH) antagonists such as leuprolide or goserelin (patients must remain on LHRH analogue therapy for the duration of the study if not surgically castrated). Progressive disease should be documented by:

  a. PSA progression (defined as two consecutive increases in PSA over a previous reference value, with the first increase in PSA occurring at a minimum of 1 week after the reference value [obtained within 2 months prior to study randomization] and confirmed by a subsequent increase in PSA whose value must be ³ 5 ng/mL prior to study randomization);41 and one of the following: i. Bone metastases (defined as ³3 foci on bone scan and confirmed radiologically within 1 month prior to study randomization); or ii. Measurable non-bony metastatic disease (documented by radiographic studies performed within 1 month prior to study randomization).
* Serum testosterone levels <50 ng/dL documented in non-surgically castrated patients within 21 days prior to randomization.
* Prior treatment with nonsteroidal antiandrogens (e.g., flutamide or bicalutamide) is allowed provided:
* There is evidence of disease progression (defined in Inclusion Criteria #2) following withdrawal of antiandrogens; and b. At least 4 weeks for flutamide or 6 weeks for bicalutamide have passed since last treatment.
* Prior treatment with ketoconazole and/or steroids is allowed provided at least 4 weeks have passed since last treatment. There are no restrictions for use of prednisone (5 mg twice daily) or another functionally equivalent oral corticosteroid for treatment of pain.
* In the rare instance a patient is potent, he must agree to practice an effective method of contraception including condom or abstinence, unless his sexual partner is sterile, from the time of first administration of MEDI-522 or docetaxel through 30 days after the last dose of either docetaxel or MEDI-522, whichever is the last drug discontinued.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 documented within 21 days prior to randomization.
* Life expectancy, in the opinion of the investigator, of at least 6 months.
* White blood cell (WBC) count ≥ 3,000/mm3; absolute neutrophil count (ANC) ≥ 1,500/mm3; platelet count ≥ 100,000/mm3; and hemoglobin ³ 9 g/dL documented within 21 days prior to randomization.
* Bilirubin ≤ ULN; aspartate transaminase (AST)/alanine transaminase (ALT) £1.5 times ULN or if AST/ALT is >1.5 times ULN, then alkaline phosphatase must be £2.5 times ULN; serum creatinine ≤ 1.5 mg/dL; INR within normal range, unless a patient is receiving anticoagulation therapy; and corrected serum calcium between 8.0-11.5 mg/dL documented within 21 days prior to randomization.
* Patients who had prior major surgery are eligible if at least 4 weeks have passed since their surgery and all surgical wounds have healed prior to study randomization.
* Prior radiotherapy including therapeutic isotopes is allowed provided measurable or evaluable disease that is clearly progressing is present and all acute radiation-related toxicities have resolved prior to study randomization.
* Prior treatment with unconventional therapy for malignancy (e.g., vitamins, St. John's Wort, PC-SPES, saw palmetto, or other herbal remedies) is allowed provided at least 4 weeks have passed since last treatment prior to randomization.
* Written informed consent and HIPAA authorization (USA sites only) obtained from the patient prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

* Prior chemotherapy for metastatic prostate cancer (prior adjuvant chemotherapy is allowed provided it is non-taxane based and at least 6 months have passed since last treatment).
* Prior treatment with other investigational agents within 4 weeks prior to randomization.
* Planned concurrent treatment with unconventional therapy for malignancy (e.g., vitamins, St. John's Wort, PC-SPES, saw palmetto, or other herbal other herbal remedies) based on medical history. Currently requiring anticoagulation (excluding use of heparin flush solutions for maintenance of catheter lines) for any thromboembolic disease based on medical history and physical examination.
* Current or planned participation (from the time of randomization through 30 days after the last dose of either docetaxel or MEDI-522, whichever is the last drug discontinued) in a research protocol in which an investigational agent or therapy may be administered.
* Any evidence of or history elicited by the investigator of prior treatment with MEDI-522 or MEDI-523.
* Prior treatment with calcitonin, mithramycin, or gallium nitrate within 2 weeks prior to randomization.
* Clinically evident central nervous system (CNS) metastasis.
* History of prior malignancies within the past 5 years other than adequately treated basal cell or squamous cell skin cancer or Stage I or II cancer currently in complete remission;
* Any evidence of or history elicited by the investigator of symptomatic cerebrovascular events (i.e., stroke or transient ischemic attack) within 6 months prior to randomization; or any history or evidence of pulmonary embolism or thrombophlebitis (including deep vein thrombosis) requiring anticoagulant therapy (e.g., warfarin or heparin).
* Any evidence of or history elicited by the investigator of myocardial infarction or angina within 6 months prior to randomization.
* Any evidence of or history elicited by the investigator of hematemesis, melena, hematochezia, or uncontrolled gross hematuria within 4 weeks prior to randomization.
* Any evidence of or history elicited by the investigator of bleeding diatheses.
* Major elective surgery planned from the time of randomization through 30 days after the last dose of either docetaxel or MEDI-522, whichever is the last drug discontinued.
* Any evidence of or history elicited by the investigator of hypersensitivity to a previously administered monoclonal antibody.
* Any evidence of or history elicited by the investigator of hypersensitivity to drugs formulated with polysorbate 80, prednisone (or other functionally equivalent oral corticosteroid), or zoledronic acid.
* Known human immunodeficiency virus (HIV) or known active viral hepatic infections based on medical history and physical examination.
* Any evidence of or history elicited by the investigator of uncontrolled or refractory hypertension or uncontrolled diabetes despite medication within 6 months prior to randomization.
* Any evidence of or history elicited by the investigator of an active infection requiring parenteral anti-infective therapy.
* A general medical or psychological condition or behavior, including substance dependence or abuse that, in the opinion of the investigator, might not permit the patient to complete the study or sign the informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-12; Primary Completion 2007-04 (Estimated); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | Baseline to disease progression
PSA Response Rate | Baseline to disease progression
Tumor Response Rate | Baseline to disease progression

SECONDARY OUTCOMES:
Anti-bone resorption assessed as the incidence of skeletal related events (SREs). (SREs) are defined as radiotherapy, surgery, pathologic bone fracture, spinal cord fracture. Overall survival will also be measured. | Baseline to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Luz Hammershaimb, MD, Study Director — MedImmune LLC
Locations (57):
- United States (36):
  - Clinical Research Consultants, Inc., Hoover, Alabama
  - Highlands Oncology Group, P.A., Springdale, Arizona
  - Arizona Hematology-Oncology, P.C., Tucson, Arizona
  - South Valley Medical Plaza, Gilroy, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Saint Francis Memorial Hospital, San Francisco, California
  - Stanford Advanced Medical Center, Stanford, California
  - Florida Cancer Specialist, Fort Myers, Florida
  - The Florida Wellcare Alliance, L.C., Inverness, Florida
  - Hemotology/Oncology Associates, Lake Worth, Florida
  - Hawaii Medical Consultants, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Ingalls Hospital, Harvey, Illinois
  - The Community Hospital, Munster, Indiana
  - Hematology Oncology Services, LLC, New Orleans, Louisiana
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - North Mississippi Hematology & Oncology Associates, Ltd., Tupelo, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - New Mexico Oncology Hematology, Consultants Ltd., Albuquerque, New Mexico
  - SUNY Down State Medical Center, Brooklyn, New York
  - VA Western New York Healthcare System, Buffalo, New York
  - North Shore Hematology Oncology Assoc., PC, East Setauket, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - VA Medical Center, Northport, New York
  - Raleigh Hematology Oncology Association, Raleigh, North Carolina
  - Clinical Research Services, Bismarck, North Dakota
  - University of Cincinnati, Barrett Cancer Center, Cincinnati, Ohio
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - Danville Hematology and Oncology, Danville, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Western Washington Oncology, Inc., P.S., Lacey, Washington
- Belgium (4):
  - A.Z. Middelheim, Antwerp
  - University Hospital Erasme, Brussels
  - Az Groeninge, Kortrijk
  - H.-Hartziekenhuis Medische Onocology-Hematologie, Roeselare
- Centre Hospitalier de L'Universite de Montreal, Montreal, Canada
- Hungary (2):
  - Borsod County Teaching Hospital, Miskolc, H
  - Szolnoki Mav Hospital, Szolnok
- Israel (3):
  - Sapir Medical Center - Meir Hospital, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Samodzielny Publiczny Wojewodzki Szpital Zespolony, Słupsk, Poland
- Russia (10):
  - Arkhangelsk Regional Oncology Center, Arkhangelsk
  - Chelyabinsk Regional Oncology Center, Chelyabinsk
  - Kazan City Oncology Center, Kazan'
  - Blokhin Cancer Research Center, Moscow
  - Russian Research Center of Radiology, Moscow
  - Semashko Central Clinical Hospital, Moscow
  - Medical Rediological Research Centre of Ran, Obninsk
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Samara Regional Oncology Center, Samara
  - Voronezh Regional Oncology Clinical Center, Voronezh